CLINICAL TRIAL: NCT00182000
Title: A Randomized, Double-Blind, Placebo-Controlled Medication Trial With D-Cycloserine for Individuals With OCD Currently Receiving Behavior Therapy
Brief Title: Effectiveness of D-Cycloserine as an Aid to Enhance Learning for Individuals With OCD Receiving Behavior Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, Director, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003-P-001325
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cycloserine; Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Seromycin (Active Comparator)
  Interventions: Drug: seromycin; Behavioral: Behavior Therapy
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Behavior Therapy

INTERVENTIONS:
Drug: seromycin — 100mg tablet administered 1 hour prior to each therapy session
  Other Names: D-Cycloserine
  Arms: Seromycin
Behavioral: Behavior Therapy — 10 weekly hour-long behavior therapy sessions

SUMMARY:
This study will assess the effectiveness of Seromycin (D-cycloserine) in enhancing the positive effects of behavior therapy for people with Obsessive-Compulsive Disorder (OCD).

DETAILED DESCRIPTION:
We hope to enroll 50 subjects in a double-blind, placebo-controlled study of D-cycloserine augmentation of behavior therapy for Obsessive-Compulsive Disorder. All subjects will undergo a pre-treatment assessment, and then be randomly assigned to receive Seromycin (100 mg) or placebo one-hour before each of 10 therapy sessions. Subjects will then come in for a treatment planning session and the behavior therapy sessions delivered twice weekly for 5 weeks. Comprehensive assessments of obsessive-compulsive symptoms, mood state, and cognitions will be given at baseline, after 5 treatment sessions, after 10 sessions and 1 month and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Structured Clinical Interview for DSM-IV (SCID) diagnosis of Obsessive Compulsive Disorder
* Score of greater than 16 on the Yale-Brown Obsessive Compulsive Scale
* Negative urinary beta-Human Chorionic Gonadotropin (hCG) test

Exclusion Criteria:

* Currently taking or have taken an unstable dose of psychotropic medications within 2 months prior to enrollment
* Currently taking medications that may interfere with the study medication
* History of seizure disorder or other serious medical illnesses (e.g., cardiovascular, liver, kidney, respiratory, endocrine, neurologic, or blood-related disease)
* Current diagnosis of tuberculosis
* Other psychiatric diagnoses (e.g., alcohol dependence, bipolar disorder, psychosis, organic mental disorder, or development disorder) that are of greater concern than the obsessive-compulsive disorder diagnosis
* Currently taking medications that may lower seizure threshold (e.g., including clozapine, pethidine, and the following antibiotics in high dosage: penicillins, cephalosporins, amphotericin, and imipenem)
* Poses a serious suicidal or homicidal threat
* Currently undergoing psychotherapy
* Failure to benefit from ten or more sessions of previous Exposure and Response Prevention (ERP) treatment
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-11; Primary Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, Ph.D., Principal Investigator — Massachusetts General Hospital

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 participants enrolled in the study. However, 4 participants decided not to participate in between consenting and starting treatment.
Groups:
- Seromycin: 10 twice-weekly sessions of behavior therapy plus 100mg tablet of seromycin
- Placebo: 10 twice-weekly sessions of behavior therapy plus 100mg tablet of placebo
Period: Overall Study
Arm/Group | Seromycin | Placebo
Started | 14 | 15
Completed | 9 | 13
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Seromycin | Placebo | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.29 (13.01) | 38.07 (12.28) | 38.18 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Yale-Brown Obsessive Compulsive Scale (YBOCS)
Description: A clinician-rated measure of obsessive-compulsive disorder severity. Each item is scored on a 0 to 4 range. Total scores are obtained by summing items 1-10 and thus range from 0 to 40 with higher scores indicating greater symptom severity. Results posted below are from the post-treatment evaluation (after 10 treatment sessions).
Time Frame: Post-treatment (week 5)
Population: Thirty-three participants were enrolled. Four participants decided not to participate in between enrolling and beginning treatment. Six participants withdrew from the study before the mid-treatment evaluation; 1 participant withdrew from the study after the mid-treatment evaluation, and this participant's data was carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Seromycin | Placebo
Number analyzed (Participants) | 10 | 13
units on a scale | 10.2 (7.2) | 14.5 (6.4)

2. Secondary Outcome: Clinical Global Impressions Scale (CGI)
Time Frame: Post-treatment (week 5)
Reporting Status: Not Posted

3. Secondary Outcome: Beck Depression Inventory (BDI)
Time Frame: Post-treatment (week 5)
Reporting Status: Not Posted

4. Secondary Outcome: Beck Anxiety Inventory (BAI)
Time Frame: Post-treatment (week 5)
Reporting Status: Not Posted

5. Secondary Outcome: Obsessional Beliefs Questionnaire (OBQ)
Time Frame: Post-treatment (week 5)
Reporting Status: Not Posted

6. Secondary Outcome: Short-Form Health Survey (SF-36)
Time Frame: Post-treatment (week 5)
Reporting Status: Not Posted

7. Secondary Outcome: Disability Inventory
Time Frame: Post-treatment (week 5)
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Seromycin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes